CLINICAL TRIAL: NCT01793974
Title: A Study of the Genetic Causes of Latent Autoimmune Diabetes in Adults
Brief Title: Genetics of Latent Autoimmune Diabetes in Adults
Acronym: LADA
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 11-008065
Record Dates: First submitted 2013-02-04; First posted 2013-02-18 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Latent Autoimmune Diabetes in Adult
Keywords: LADA; Latent Autoimmune Diabetes in Adults; Latent Autoimmune Diabetes; Latent Diabetes in Adults
MeSH Terms: conditions — Latent Autoimmune Diabetes in Adults

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Latent Autoimmune Diabetes in Adult: Individuals who meet criteria for Latent Autoimmune Diabetes in Adult
- Without Latent Autoimmune Diabetes in Adult: Individuals who do not meet criteria for Latent Autoimmune Diabetes in Adult

SUMMARY:
This is a prospective study that will study adults and has the objective of examining 'Latent Autoimmune Diabetes in Adults' (LADA) to understand how this trait is influenced by genetic factors.

DETAILED DESCRIPTION:
A case-control study approach will be used to compare the allelic frequencies of Deoxyribonucleic acid (DNA) markers of the cases (i.e., LADA patients) to a randomly selected control samples that does not have the trait under study. To study the role of genetic factors in LADA, the study seeks to determine if certain genomic regions that are captured or mirrored by selective Single nucleotide polymorphisms (SNPs) that are genotyped, are over or underrepresented in those with the disease compared to those who do not. The level of auto-antibodies is the serum can also be studied as a quantitative trait where we ask the question if there is correlation with specific SNP alleles that are genotyped. The markers that are found to be over or under-represented in the study cases will then be tested in an independent set of patients also recruited in this study. This allows us to filter markers that show significance simply by chance and prevents us from being misled.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed type 2 Diabetes (T2D) patient with: BMI <30 at diagnosis; Age >25-<50 at diagnosis

OR

* Diagnosed type 1 Diabetes (T1D) patient with: Age >25 at diagnosis

OR

- Currently Diagnosed with LADA with age at initial diagnosis of Diabetes >25 years and a positive GAD65 antibody test

Exclusion Criteria:

* Any underlying disease or condition that is a contraindication for obtaining 18.0 ml of blood.
* Inability to obtain an informed consent from a given LADA case.
* Blood sampling has already occurred for a given subject.
* Previous GAD65 antibody test(s) negative.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment will be carried out at several adult diabetes clinics across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2011-07; Primary Completion 2015-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Identify variations in the human genome associated with LADA by genotyping cases and comparing allele frequencies to an existing control database | 5 years

SECONDARY OUTCOMES:
Identify associations between genetic variants with certain measurable risk profiles that can be used to judge the health status or well being of a LADA case. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Struan Grant, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States
- The University of Leicester, Leicester, United Kingdom